CLINICAL TRIAL: NCT04850092
Title: Investigation on Dynamic Arterial Elastance as a Predictor of Hypotension Caused by the Positional Change From Supine to Prone (SuProne Study).
Brief Title: Dynamic Arterial Elastance to Predict Postural Change Induced Hypotension
Status: Completed | Type: Observational
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Eunah Cho, MD, Assistant Professor, Kangbuk Samsung Hospital
Other Study IDs: KBSMC 2021-04-038
Record Dates: First submitted 2021-04-14; First posted 2021-04-20 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-hypotensive: Mean blood pressure is maintained after positional change from supine to prone.
  Interventions: Other: Positional change from supine to prone
- Hypotensive: Mean blood pressure decrease < 20% after positional change from supine to prone.
  Interventions: Other: Positional change from supine to prone

INTERVENTIONS:
Other: Positional change from supine to prone — Patient is turned from supine to prone position for spine surgery

SUMMARY:
During general anesthesia, hypotension might occur during positional change. It is reported that hypotension after positional change from supine to prone is mainly caused by the decrease in preload. The investigators aimed to investigate whether dynamic arterial elastance might predict hypotension associated with positional change from supine to prone.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for invasive arterial catheter insertion, undergoing elective spine surgery in prone position under general anesthesia

Exclusion Criteria:

* arrythmia
* pulmonary disease
* increased intracranial pressure
* decreased cardiac function (ejection fraction < 50%)
* obesity (body mass index > 40)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are scheduled for spine surgery and need positional change from supine to prone positioin.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Dynamic arterial elastance before positional change | 1 minute before positional change
  Dynamic arterial elastance, defined as the ratio of pulse pressure variance/stroke volume variance will be recorded 1 minute before positional change

CONTACTS AND LOCATIONS:
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided